CLINICAL TRIAL: NCT07201532
Title: Disease Modification Outcomes in Diabetes: a Delphi Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Other Study IDs: 4602UE
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare practitioners and researchers: Healthcare practitioners and researchers working in the field of diabetes research and/or clinical care
  Interventions: Other: eDelphi method
- People with type 2 diabetes
  Interventions: Other: eDelphi method

INTERVENTIONS:
Other: eDelphi method — A Delphi consensus study will be undertaken to establish a core outcome set for disease modification in type 2 diabetes.

SUMMARY:
Type 2 diabetes is a condition when the pancreas does not produce enough of the hormone, insulin, or the insulin that is formed does not function effectively. This results in high blood sugar levels. Type 2 diabetes is associated with other health conditions, and people with the condition have a higher chance of dying earlier and having other complications. People with type 2 diabetes take a lot of different types of medications. The current treatments that exist aim to manage blood sugar levels, rather than affect the progression of the disease.

The research involving treatments that impact the long-term progression of type 2 diabetes is sometimes hard to understand. This is because research studies measure a lot of different outcomes (outcomes are items we measure to show that the study has worked and/or it is safe). One way of improving research is to make sure that we are measuring the same outcomes, but also that these outcomes are important to people living with type 2 diabetes and healthcare professionals. This can be done by using a core outcome set (COS). A COS is a short list of outcomes that are important to researchers, healthcare professionals and people living with type 2 diabetes. The aim of this study is to design a COS for research studies for disease modification in type 2 diabetes via an e-Delphi study.

The Delphi process is a structured process used for forming a consensus, where stakeholder groups provider their opinions in an iterative approach for answering questions over several rounds. This will also take place using surveys online.

ELIGIBILITY:
Inclusion Criteria:

Participants will fall into one of two groups:

1. Healthcare practitioners and researchers working in the field of diabetes research and/or clinical care.
2. People with type 2 diabetes. All participants will be ≥18 years of age.

Exclusion Criteria:

1. Potential participants who are not willing to provide informed consent or participate in the Delphi study.
2. Those who are unable to understand English.
3. Those without the capability to respond to the online survey.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthcare practitioners and researchers working in the field of diabetes research and/or clinical care and people with type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Delphi Round 1 | Three to four weeks
  The Delphi methodology is an interactive multi-stage process, with each stage building on the data of the previous results in order to gain consensus from the participants. This is achieved through a series of surveys interspersed with controlled feedback containing the aggregated results from all participants in the study cohort.
  In Delphi Round 1, participants will be asked to rate the importance of outcomes for inclusion or exclusion using a 9-point Likert scale.
Delphi Round 2 | Three to four weeks
  In Round 2, participants will be asked to rate the importance of remaining outcomes that did not reach consensus for inclusion or exclusion in Round 1 using a 9-point Likert scale. Consensus is defined as a minimum of 70% of participants who rated an outcome as 1-3 "Not important" and should be excluded or 7-9 and indicates an outcome is "Critical" and should be included.
  If necessary, a third round of the survey will be administered to attempt to reach consensus on the remaining outcomes/instruments that did not do so in the previous rounds. Results will inform the development of the final COS.